CLINICAL TRIAL: NCT02131675
Title: Observational Study of C-peptide Levels in Youth With Longstanding Type 1 Diabetes Mellitus as Detected by an Ultrasensitive Assay
Brief Title: Detection of C-peptide in Youth With Longstanding Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-1425
Record Dates: First submitted 2014-04-08; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: C-peptide; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Boost shake: children that have had type 1 diabetes for more than 1 year
  Interventions: Dietary Supplement: Boost shake

INTERVENTIONS:
Dietary Supplement: Boost shake — Blood draw after mixed-meal consumption
  Other Names: mixed-meal

SUMMARY:
Background Type 1 diabetes is characterized by pancreatic beta-cell destruction and an inability to synthesize insulin. Connecting peptide (C-peptide) is formed from the same precursor as insulin and is produced in equimolar amounts as insulin. There are several clinical trials currently being performed to explore the possibility of beta-cell preservation or regeneration. Most children are not eligible for these trials because it is often presumed that C-peptide levels will decrease and become undetectable after years of having type 1 diabetes. Several studies in the adult population have demonstrated that C-peptide may remain measureable in patients who have had diabetes for up to 50 years after diagnosis. Recently, it was demonstrated that 10% of adult patients who have had type 1 diabetes for 31-40 years have measureable levels of serum C-peptide if measured with an ultrasensitive assay. The levels were lower in patients who had diabetes for a longer time. This pattern was also demonstrated in the Diabetes Control and Complications Trial (DCCT) and NHANES trial. No studies have been performed exclusively in pediatric patients Hypothesis The investigators hypothesize that C-peptide should be detectable in the sera of pediatric patients who have had type 1 diabetes for greater than 1 year and as far out as > 20 years after diagnosis. The investigators also hypothesize that since their patient population has had diabetes for less time as compared to adults, the levels of C-peptide should be higher than reported for adults and that a greater proportion of patients in the pediatric population will have detectable C-peptide levels as compared to adults.

DETAILED DESCRIPTION:
1) Objectives:

1. To determine if C-peptide is detectable in the sera of children that have had type 1 diabetes for more than 1 year using an ultrasensitive assay.
2. To correlate C-peptide levels with duration since diagnosis, current age, antibody titers at diagnosis, hemoglobin A1c, total daily insulin dosage.
3. To determine responsiveness of residual C-peptide to mixed-meal testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 1-25 years of age
* Have had type 1 diabetes for more than 1 year.

Exclusion Criteria:

* Does not meet inclusion criteria
* Foster children
* Patients without primary caregiver
* Pregnant

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the population of patients seen in the Division of Pediatric Endocrinology and Diabetes. These patients must have type 1 diabetes and must have been diagnosed more than 1 year prior to their recruitment. Potential subjects will be identified by reaching out to the physicians in the division and asking that they inform the investigators of patients that they see with type 1 diabetes. Those patients will have their information reviewed by the investigators using EPIC, the electronic medical record at The Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
C-peptide level | Day 1

SECONDARY OUTCOMES:
Hemoglobin A1c | Day 1
  Hemoglobin A1c at diabetes diagnosis and at most recent medical visit will be correlated with C-peptide level
Total daily dose of insulin | Day 1
  Total daily dose of insulin per kilogram will be correlated with C-peptide level
Age at diabetes diagnosis | Day 1
  Age at diabetes diagnosis will be correlated with C-peptide level
Duration of diabetes | Day 1
  Duration of diabetes will be correlated with C-peptide level

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rapaport, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Evan Graber, DO, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Sperling MA, Weinzimer SA, Tamborlane WV. Diabetes Mellitus. In: Sperling MA ed. Pediatric Endocrinology. 3rd ed. Philadelphia, PA: Saunders Elsevier; 2008:385
- [Background] Wherrett DK, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Herold KC, Marks JB, Monzavi R, Moran A, Orban T, Palmer JP, Raskin P, Rodriguez H, Schatz D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet GAD Study Group. Antigen-based therapy with glutamic acid decarboxylase (GAD) vaccine in patients with recent-onset type 1 diabetes: a randomised double-blind trial. Lancet. 2011 Jul 23;378(9788):319-27. doi: 10.1016/S0140-6736(11)60895-7. Epub 2011 Jun 27. PMID 21714999
- [Background] Orban T, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Marks JB, Monzavi R, Moran A, Raskin P, Rodriguez H, Russell WE, Schatz D, Wherrett D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Abatacept Study Group. Co-stimulation modulation with abatacept in patients with recent-onset type 1 diabetes: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jul 30;378(9789):412-9. doi: 10.1016/S0140-6736(11)60886-6. Epub 2011 Jun 28. PMID 21719096
- [Background] Pescovitz MD, Greenbaum CJ, Krause-Steinrauf H, Becker DJ, Gitelman SE, Goland R, Gottlieb PA, Marks JB, McGee PF, Moran AM, Raskin P, Rodriguez H, Schatz DA, Wherrett D, Wilson DM, Lachin JM, Skyler JS; Type 1 Diabetes TrialNet Anti-CD20 Study Group. Rituximab, B-lymphocyte depletion, and preservation of beta-cell function. N Engl J Med. 2009 Nov 26;361(22):2143-52. doi: 10.1056/NEJMoa0904452. PMID 19940299
- [Background] Gottlieb PA, Quinlan S, Krause-Steinrauf H, Greenbaum CJ, Wilson DM, Rodriguez H, Schatz DA, Moran AM, Lachin JM, Skyler JS; Type 1 Diabetes TrialNet MMF/DZB Study Group. Failure to preserve beta-cell function with mycophenolate mofetil and daclizumab combined therapy in patients with new- onset type 1 diabetes. Diabetes Care. 2010 Apr;33(4):826-32. doi: 10.2337/dc09-1349. Epub 2010 Jan 12. PMID 20067954
- [Background] Wang L, Lovejoy NF, Faustman DL. Persistence of prolonged C-peptide production in type 1 diabetes as measured with an ultrasensitive C-peptide assay. Diabetes Care. 2012 Mar;35(3):465-70. doi: 10.2337/dc11-1236. PMID 22355018
- [Background] Keenan HA, Sun JK, Levine J, Doria A, Aiello LP, Eisenbarth G, Bonner-Weir S, King GL. Residual insulin production and pancreatic ss-cell turnover after 50 years of diabetes: Joslin Medalist Study. Diabetes. 2010 Nov;59(11):2846-53. doi: 10.2337/db10-0676. Epub 2010 Aug 10. PMID 20699420
- [Background] Effects of age, duration and treatment of insulin-dependent diabetes mellitus on residual beta-cell function: observations during eligibility testing for the Diabetes Control and Complications Trial (DCCT). The DCCT Research Group. J Clin Endocrinol Metab. 1987 Jul;65(1):30-6. doi: 10.1210/jcem-65-1-30. PMID 2884229
- [Background] Greenbaum CJ, Anderson AM, Dolan LM, Mayer-Davis EJ, Dabelea D, Imperatore G, Marcovina S, Pihoker C; SEARCH Study Group. Preservation of beta-cell function in autoantibody-positive youth with diabetes. Diabetes Care. 2009 Oct;32(10):1839-44. doi: 10.2337/dc08-2326. Epub 2009 Jul 8. PMID 19587365